CLINICAL TRIAL: NCT03224741
Title: Behavioral Nudges, Information and Incentives for HIV Testing: A Field Experiment in Ecuador
Brief Title: Behavioral Economics Field Experiment in HIV Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Universidad San Francisco de Quito (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: HIRB00004772
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: HIV/AIDS Serodiagnosis
Keywords: Behavioral Economics

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: The subject receives the script and actions associated with the experimental condition she/he is assigned to according to the randomization. The subject receives a card consisting of three detachable parts. Each part includes a numerical ID that uniquely identifies each participant. The first part of the card will remain with the researchers. The second part of the card does to the medical personnel at the health facility if and when they go there to get tested. The third part of the card will remain with the participant. This procedure and the study ID will enable the research team to (a) associate participants to the treatment conditions and (b) determine the outcomes (whether they got tested or not, and what the results were), while preserving the anonymity of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Information (Placebo Comparator)
  Interventions: Behavioral: Information
- Active Choice (Active Comparator)
  Interventions: Behavioral: Active Choice
- Monetary incentive (Experimental)
  Interventions: Behavioral: Monetary Incentive

INTERVENTIONS:
Behavioral: Monetary Incentive — Subjects in this condition will be read a script informing them of the benefits and importance of routine HIV/AIDS testing for themselves, the benefits for one's partner and loved ones, and for the broader community; they are also given a flyer including the same information.Iin addition, they will be told that if they will get tested for HIV/AIDS within the next two weeks, they will receive $10 (the US dollar became Ecuador's official currency in 2001).
  Arms: Monetary incentive
Behavioral: Information — Subjects assigned to this condition are read a script informing them of the benefits and importance of routine HIV/AIDS testing for themselves, the benefits for one's partner and loved ones, and for the broader community; they are also given a flyer including the same information. Then, they are invited to get tested in the next two weeks.
  Arms: Information
Behavioral: Active Choice — Subjects in this condition will receive the same information and flyer as in T1; in addition, they are told that they have the opportunity to express their intention to get tested for HIV/AIDS. To this aim, they will be given a sheet of paper and asked to tick one of two boxes. The first box will say "I intend to get tested within the next two weeks", and the second will say "I will consider getting tested within the next two weeks but I am not ready to commit at this time". They will also be asked to write their initials at the bottom of the sheet, and will be told to keep it. This is a form of "soft commitment" which has proven effective in other contexts (Bryan et al. 2010).
  Arms: Active Choice

SUMMARY:
The investigators propose to conduct a randomized controlled trial in collaboration with the Fundacion Raices, a non-governmental organization (NGO) with strong ties to the local community of Esmeraldas, Ecuador. A total of about 3,000 subjects will be involved in the full-scale study over the course of 2 years. In partnership with the Fundacion Raices, the research team will set up stands at four public places in the city of Esmeraldas: the "malecon" (esplanade on the town's waterfront), the "Centro Comercial Multiplaza" (Esmeraldas' large shopping mall), the municipal market (a popular destination for groceries, etc.), and a public park located in the city center. Each stand will feature a sign inviting individuals to stop and "get their health checked", and will provide free refreshments (juice boxes and water). A monitor will approach individuals at the malecon/shopping center/municipal market/public park and ask whether they are interested to learn about a health initiative by the Fundacion Raices and a group of public health researchers. If an individual is interested, the monitor will begin the three steps of the experiment:

1. Participants fill out a brief, anonymous survey with demographics, socio- economic characteristics, and whether they have been tested for HIV/AIDS in the past.
2. Participants receive the script and actions associated with the experimental condition into which they are assigned to according to the randomization table.

   There are three experimental conditions:

   T1 = "Information". T2 = "Active Choice". T3 = "Monetary incentive".
3. Whether participants subsequently showed up at a medical facility to get tested for HIV/AIDS is noted in the record.

DETAILED DESCRIPTION:
The investigators propose to conduct a randomized controlled trial in collaboration with the Fundacion Raices, a non-governmental organization (NGO) with strong ties to the local community of Esmeraldas, Ecuador. A total of about 3,000 subjects will be involved in the full-scale study over the course of 2 years. In partnership with the Fundacion Raices, the research team will set up stands at four public places in the city of Esmeraldas: the "malecon" (esplanade on the town's waterfront), the "Centro Comercial Multiplaza" (Esmeraldas' large shopping mall), the municipal market (a popular destination for groceries, etc.), and a public park located in the city center. Each stand will feature a sign inviting individuals to stop and "get their health checked", and will provide free refreshments (juice boxes and water). A monitor will approach individuals at the malecon/shopping center/municipal market/public park and ask whether they are interested to learn about a health initiative by the Fundacion Raices and a group of public health researchers. If an individual expresses interest, a field worker will begin the three steps of the experiment: (1) The participant completes a brief, anonymous survey with demographics, socio- economic, and past HIV/AIDS testing information. (2) The participant receives the script and actions associated with the assigned randomized experimental condition. There are three experimental conditions: - T1 = "Information". T2 = "Active Choice". T3 = "Monetary incentive". (3) Whether the participant shows up at the medical facility to get tested is entered in the record.

Randomization: The randomization will vary by week (i.e., all participants who present on the same week will be assigned to the same experimental condition) to minimize spillover effects due to communication between participants assigned to different groups, and to avoid confusion among the field staff.

The implementation schedule will be designed to guarantee balance of treatment conditions across locations and days of the week. To provide the participants with privacy when filling the questionnaire, after the initial approach, the interaction between the participants and field staff will occur in a booth next to the desk which will obscure the participant from the view of others. Participants will be read a statement inviting participation; description of privacy protection measures; and solicitation of verbal consent.

The investigators also plan to test our experimental conditions with subjects from high-risk population groups. For high-risk population groups, the investigators will rely on the previous experience of research team members in which Female Sex Workers (FSWs) and Men who have Sex with Men (MSM) were contacted through the official registry and local MSM association, respectively. A similar approach will be used in this project. Participants in these high-risk groups will be approached individually by field staff, after having been randomly assigned to one of three experimental conditions. Participants will be read a statement inviting participation; description of privacy protection measures; and solicitation of verbal consent. The investigators expect to include about 1,000 subjects from the high-risk populations.

The medical testing facility where participants will go is "Microlab - Laboratiorio Clinico Bacteriologico", centrally located in Esmeraldas (across the street from the Delfina Torres Public Hospital). It is a private facility staffed by healthcare professionals connected to the testing lab at the Medical School and Hospital of the Universidad San Francisco de Quito (USFQ) in Quito, Ecuador. Blood samples will be tested using standardized commercially available HIV testing kits. Participants in the financial incentive condition will receive their reward from the staff at the Microlab in Esmeraldas. The participants will not provide names to the lab personnel. Instead, they will give them the second portion of the registration card, which indicates their study identification number (ID). The lab staff will write the study ID onto the sample collection label. Blood samples will be sent to the testing facility at the USFQ. There, trained laboratory personnel will conduct the HIV screening test following Standard Operating Procedures. After conducting the test, laboratory personnel will record the results in an excel spreadsheet using the participant's ID number as identifier (i.e., there will be no record of name or other personal identifiable information).

Afterwards, the results will be individually printed on a pre-designed "HIV screening Test Results" Form. Individual results will be put in an envelope. Envelopes will be sealed and sent back to the testing facility in Esmeraldas via a private carrier. After arrival, results will be archived in a locked unit and delivered to participants as they arrive to claim their results. Participants will receive their results in a timely manner, according to local health policies. HIV positive individuals will be encouraged to visit the local health district to enroll into the national HIV/AIDS program for treatment.

ELIGIBILITY:
Inclusion Criteria:

* All participants able to understand the instructions and provide consent

Exclusion Criteria:

* Under 18 years of age (age of consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7720 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in each experimental condition that showed up for the HIV sero test. | 2 weeks
  The outcome measure is a relative proportion of participants in each experimental condition that showed up at the 'Microlab - Laboratiorio Clinico Bacteriologico' to provide a blood sample for the HIV sero test. It is calculated as the number of tested participants divided by the total number of participants enrolled into each experimental condition. An enrolled participant is defined as an individual that received the information and instructions in T1, T2 and T3.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Francisco de Quito, Quito, Ecuador

IPD SHARING:
Plan to Share IPD: No